CLINICAL TRIAL: NCT00000970
Title: A Phase I Open-Labeled Study of Long Term Combined or Alternating Foscarnet/Ganciclovir Maintenance Therapy for AIDS Patients With CMV Retinitis After Ganciclovir Induction Therapy
Brief Title: A Study of Foscarnet Plus Ganciclovir in the Treatment of Cytomegalovirus of the Eye in Patients With AIDS Who Have Already Been Treated With Ganciclovir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Astra USA (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 151; 11126 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Ganciclovir; Drug Evaluation; Drug Therapy, Combination; Foscarnet; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet; Ganciclovir

INTERVENTIONS:
Drug: Foscarnet sodium
Drug: Ganciclovir

SUMMARY:
To examine the safety and tolerance of the administration of ganciclovir and foscarnet given together or alternately; to determine the interactive pharmacokinetics (blood level) profile of long-term combined and alternating therapy with these two drugs. Additional objectives are to examine the effect of these treatments in controlling time to cytomegalovirus (CMV) retinitis progression and to examine the antiviral activity of combined and alternating ganciclovir/foscarnet treatment and development of antiviral resistance. Sight-threatening CMV retinitis occurs in at least 6 percent of AIDS patients. By 1991 (US), there may be 6000 to 10000 patients with CMV retinitis. Many clinical reports suggest that both ganciclovir (DHPG) and foscarnet have an antiviral effect against CMV that is often associated with clinical stabilization. Effectiveness of ganciclovir and foscarnet is correlated with weekly maintenance and since toxicity is dose-limiting in up to 20 percent of patients receiving either drug for long periods, it may be beneficial in long-term maintenance treatment to combine or alternate these two drugs at a lower total weekly dose of each drug.

This strategy may result in a greater net antiviral effect with less toxicity than is seen with either drug alone, because the toxicities of each drug are quite different.

DETAILED DESCRIPTION:
Sight-threatening CMV retinitis occurs in at least 6 percent of AIDS patients. By 1991 (US), there may be 6000 to 10000 patients with CMV retinitis. Many clinical reports suggest that both ganciclovir (DHPG) and foscarnet have an antiviral effect against CMV that is often associated with clinical stabilization. Effectiveness of ganciclovir and foscarnet is correlated with weekly maintenance and since toxicity is dose-limiting in up to 20 percent of patients receiving either drug for long periods, it may be beneficial in long-term maintenance treatment to combine or alternate these two drugs at a lower total weekly dose of each drug.

This strategy may result in a greater net antiviral effect with less toxicity than is seen with either drug alone, because the toxicities of each drug are quite different.

All patients have newly diagnosed CMV retinitis and have completed a 14-day course of intravenous ganciclovir or foscarnet induction therapy within 1 week prior to study entry. The maintenance period consists of a 12-week study period followed by a 40 week follow-up period. Treatment consists of either combined sequential daily maintenance therapy of both foscarnet and ganciclovir or alternating daily treatment with ganciclovir one day and foscarnet the following day.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemotherapy for Kaposi's sarcoma (excluding interferon) if patient is hematologically stable for at least 30 days prior to entry.
* Zidovudine (AZT), dideoxyinosine (ddI), dideoxycytidine (ddC) after first two weeks of study period if absolute neutrophil count is > 1000 cells/mm3 and hemoglobin = or > 8 g/dl.
* Vancomycin.
* Fluconazole or investigational triazoles (e.g., itraconazole, SCH 39304) for disseminated fungal infection.
* Pneumocystis carinii pneumonia prophylaxis (except parenteral pentamidine).
* Acyclovir or other appropriate medication may be instituted in the event of the appearance of Herpes simplex virus
* (HSV) or Varicella zoster virus (VZV) infections.
* G-CSF or GM-CSF for grade 4 neutropenia.

Concurrent Treatment:

Allowed:

* Recombinant human erythropoietin.

Prior Medication: Required:

* Completion of 14-day course of intravenous ganciclovir induction therapy (2.5 mg/kg IV q8h or 5 mg/kg q12h for 14 days) or foscarnet induction therapy (60 mg/kg q8h adjusted for renal function for 14 days) within 1 week prior to study entry. Patients who do not initiate the study immediately upon completing ganciclovir induction therapy should receive a maintenance ganciclovir regimen of 5 mg/kg/day or 6 mg/kg/day 5 x week or a foscarnet regimen of 90-120 mg/kg/day until initiating study drug.

Patients must:

* Have a diagnosis of cytomegalovirus retinitis and HIV infection.
* Be capable of giving informed consent. Patients < 18 years of age may participate with the consent of parent, guardian, or person with power of attorney.

Allowed:

* History of seizure disorder or a central nervous system (CNS) mass lesion.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Evidence of tuberculous, diabetic or hypertensive retinopathy.
* Osteomalacia, neoplasm metastatic to bone or other bone disease.
* Any clinically significant pulmonary or neurologic impairment (for example, patients who are intubated or comatose).
* Retinal detachment.
* Corneal, lens, or vitreous opacification precluding funduscopic exam.

Concurrent Medication:

Excluded:

* Immunomodulators, biologic response modifiers or investigational agents not specifically allowed.
* Aminoglycosides, amphotericin B, probenecid, parenteral pentamidine.
* Zidovudine (AZT), dideoxyinosine (ddI), dideoxycytidine (ddC) until completion of second week of maintenance therapy. ddC use is discouraged but not prohibited because of paucity of experience of this drug with ganciclovir and foscarnet.

Anti-cytomegalovirus (CMV) therapy:

* Ganciclovir, CMV hyperimmune serum/globulin, interferons, immunomodulators.
* Prophylactic antiviral therapy with acyclovir.

Patients with the following are excluded:

* Active AIDS-defining opportunistic infection requiring therapy that is currently causing nephrotoxicity or myelosuppression.
* Known hypersensitivity to either of the study therapies.

Prior Medication:

Excluded:

* Foscarnet or ganciclovir for CMV retinitis (excluding the 14-day induction period).

Prior Treatment:

Excluded:

* Cytomegalovirus (CMV) hyperimmune globulin within 14 days prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Study Completion 1993-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobson MA, Study Chair
Locations (6):
- United States (6):
  - USC CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - Washington U CRS, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Jacobson MA, Kramer F, Bassiakos Y, Hooton T, Polsky B, Geheb H, O'Donnell JJ, Walker JD, Korvick JA, van der Horst C. Randomized phase I trial of two different combination foscarnet and ganciclovir chronic maintenance therapy regimens for AIDS patients with cytomegalovirus retinitis: AIDS clinical Trials Group Protocol 151. J Infect Dis. 1994 Jul;170(1):189-93. doi: 10.1093/infdis/170.1.189. PMID 8014496
- [Background] Aweeka FT, Gambertoglio JG, Kramer F, van der Horst C, Polsky B, Jayewardene A, Lizak P, Emrick L, Tong W, Jacobson MA. Foscarnet and ganciclovir pharmacokinetics during concomitant or alternating maintenance therapy for AIDS-related cytomegalovirus retinitis. Clin Pharmacol Ther. 1995 Apr;57(4):403-12. doi: 10.1016/0009-9236(95)90209-0. PMID 7712668